CLINICAL TRIAL: NCT05361551
Title: Stereotactic Liver Ablation Assisted With Intra-Arterial CT Hepatic Arteriography and Ablation Confirmation Software Assessment (STEREOLAB)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0221; NCI-2022-03903 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Liver Ablation; Hepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liver ablation (Experimental): The ablation procedure will be performed in 1 day
  Interventions: Procedure: Liver ablation

INTERVENTIONS:
Procedure: Liver ablation — Ablation needle placement An image-guidance device be used for planning of the procedure and for placement of the ablation needle

SUMMARY:
To achieve adequate tumor treatment coverage with sufficient minimal ablation margins, several steps are required: firstly, it is critical to define tumor boundaries and extent on intra-procedural CT image; secondly, accurate planning, targeting, and confirmation of ablation probe placement within the tumor; thirdly, the use of an intra-procedural imaging assessment method to evaluate minimal ablation margins is required to define whether sufficient minimal ablation margins was obtained or if additional ablation is needed. Taking all together, those factors points to the need of having a high-precision ablation methodology for intra-procedural planning, monitoring, and ablation margin assessment. Currently, such methods are only utilized in isolation and the benefit of a combined and standardized procedure workflow is unknown. Therefore, our primary goal of this single-arm clinical trial is to investigate the technical efficacy of a high-precision liver ablation technique comprised by stereotactic-guidance, CT during hepatic arteriography-based imaging analysis, and computer-based software assessment of ablation margins for the treatment of patients referred to ablation for the treatment of primary and secondary liver cancers.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the technical efficacy and Local Tumor Progression-free survival [LTPFS] of a high-precision liver ablation technique comprised by stereotactic-guidance, CT during hepatic arteriography-based imaging analysis, and computer-based software assessment of ablation margins, for the treatment of patients with colorectal liver metastasis referred to percutaneous liver ablation.

Secondary Objectives:

To evaluate the impact of this high-precision liver ablation technique on:

1. Impact of minimally ablated margins on LTPFS
2. 3D Minimal ablation margins;
3. Adverse events;
4. Liver function;
5. Tissue properties from US elastography;
6. Contrast-media utilization and radiation exposure;
7. Overall oncological outcomes (disease-free and overall survival, and ability to provide salvage local therapy at the time of recurrence).
8. Anesthesia/procedural time
9. Response and Duration of response
10. Assessing whether ringenhancing hypervascular liver micronodules represent metastasis

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with up to 5 colorectal liver metastasis measuring up to 5 cm who are referred to percutaneous ablation;
2. Ability to completely cover the target tumor with at least a 5 mm ablation margin as determined per pre-procedure cross-sectional imaging;
3. Distance to central bile ducts > 1 cm;
4. Adequate glomerular filtration rate (GFR > 40) and no severe allergies to iodine contrast-media;
5. Ability to understand and the willingness to sign written informed consent;
6. Age > 18 years-old;
7. Performance status 0-2 (Eastern Cooperative Oncology Group Classification [ECOG]);
8. Expected survival > 12 months.

Exclusion Criteria:

1. Use of other prior or concomitant local therapy at the target tumor(s).
2. Active bacterial infection or fungal infection on the day of the ablation.
3. Platelet < 50,000/mm3.
4. INR > 1.5
5. Patients with uncorrectable coagulopathy.
6. Currently breastfeeding or pregnant (latter confirmed by serum pregnancy test).
7. Physical or psychological condition which would impair study participation.
8. ASA (American Society of Anesthesiologists) score of ≥ 4.
9. Any other loco-regional therapies at the target lesion(s).
10. Anatomical variations in the arterial-hepatic blood supply of the liver that preclude the use of CTHA imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire (EQ-5D-3L) | through study completion, an average of 1 year
  The scale is numbered from 0-100 (100 means the best health you can imagine. 0 means the worst health you can imagine)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Odisio, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Paolucci I, Albuquerque Marques Silva J, Lin YM, Fellman BM, Jones KA, Tatsui CE, Weinberg JS, Ruiz J, Tan J, Brock KK, Bale R, Odisio BC. Study Protocol STEREOLAB: Stereotactic Liver Ablation Assisted with Intra-Arterial CT Hepatic Arteriography and Ablation Confirmation Software Assessment. Cardiovasc Intervent Radiol. 2023 Dec;46(12):1748-1754. doi: 10.1007/s00270-023-03524-9. Epub 2023 Aug 10. PMID 37563313
- See also: M D Anderson Cancer Center — http://www.mdanderson.org